CLINICAL TRIAL: NCT04150861
Title: An Open-label Trial Investigating the Pharmacokinetics of FE 999049 Given as a Single Subcutaneous Dose in Gonadotropin Down-regulated Healthy Chinese Women
Brief Title: Rekovelle PK Trial in Chinese Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 000152
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Results first posted 2020-12-24 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2020-01

CONDITIONS: Infertility
Keywords: In vitro fertilisation; Controlled ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — follitropin delta; FE 999049

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Follitropin delta 12 μg (Experimental): Participants received single subcutaneous abdominal injection of Follitropin delta 12 μg on Day 1.
  Interventions: Drug: Follitropin Delta
- Follitropin delta 18 μg (Experimental): Participants received single subcutaneous abdominal injection of Follitropin delta 18 μg on Day 1.
  Interventions: Drug: Follitropin Delta
- Follitropin delta 24 μg (Experimental): Participants received single subcutaneous abdominal injection of Follitropin delta 24 μg on Day 1.
  Interventions: Drug: Follitropin Delta

INTERVENTIONS:
Drug: Follitropin Delta — Solution for Injection, subcutaneous administration
  Other Names: REKOVELLE; FE 999049

SUMMARY:
FE 999049 is a gonadotropin preparation containing recombinant human follicle stimulating hormone (rhFSH) under development by Ferring Pharmaceuticals. It is intended for controlled ovarian stimulation for the development of multiple follicles in women undergoing assisted reproductive technologies (ART) such as in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) cycle. In previous trials the exposure to and dose proportionality of FE 999049 in a clinically relevant dose range in Caucasian and Japanese healthy women have been shown to be very similar. This is a trial in healthy Chinese women investigating the pharmacokinetics, safety, and tolerability of a single subcutaneous dose of FE 999049.

ELIGIBILITY:
Inclusion Criteria:

* Female of Chinese origin, with two ethnic Chinese parents and four ethnic Chinese grandparents 21-40 years of age (both inclusive)
* Willing to stop using combined oral contraceptives (COC) in relation to the first DECAPEPTYL Depot administration on Day -28
* Agrees to use a double barrier method of contraception between Day -63 and Day 28, if not abstinent. A double barrier method of contraception should also be used after Day 28 until menses resumes or until another contraceptive method has been established
* Normal menstrual cycles with a range of 24-35 days in the absence of oral contraceptives
* Serum FSH less than equal to (≤)5 IU/L on Day -3 and Day -1
* Body mass index (BMI) of 18.5 -25 kg/m^2 (both inclusive)
* Negative serology for human immunodeficiency virus (HIV) antibody, hepatitis B (surface antigen), hepatitis C antibody, and syphilis bacteria
* Healthy according to medical history, physical examination, gynaecological examination, ECG, blood pressure, and laboratory profile of blood and urine
* Negative urine drug screen and alcohol breath test at screening and on Day -1
* Non-smoker or light smoker (≤ 5 cigarettes/day) for at least 6 months prior to trial

Exclusion Criteria:

* Presence or a history of clinically significant diseases of the renal, hepatic, gastrointestinal, cardiovascular, or musculoskeletal systems, or presence or history of clinically significant reproductive, psychiatric, immunological, endocrine or metabolic diseases
* Cancer within the last 5 years except for adequately managed basal cell carcinoma and squamous cell carcinoma of the skin
* Pregnancy or breastfeeding
* Current or a history of endocrine abnormalities such as hyperprolactinaemia, polycystic ovary syndrome or other ovarian dysfunction, tumours of the pituitary gland or hypothalamus, thyroid or adrenal disease
* Clinically significant findings on the trans-vaginal ultrasound, cytology, gynaecological or breast examination at screening or on Day -1 including ovarian cysts or tumours of the ovaries or uterus
* Contraindications for the use of gonadotropins and gonadotropin-releasing hormone (GnRH) agonists
* Previously treated with gonadotropins within the last 6 months prior to screening
* History within the last two years or current abuse of alcohol or drugs
* Presence or history of severe allergy or anaphylactic reactions
* Intake of prescribed medication, over-the-counter (OTC) medication, or herbal medicines, with the exceptions of COC, cromoglycate, and paracetamol according to the labelling, within 2 weeks or 5 half-lives of the drug, whichever is longer, prior to first dose of DECAPEPTYL Depot. Topical treatments of bacterial or fungal infection are allowed if stopped before first dose of IMP
* Intake of any non-registered investigational drug within the last 12 weeks preceding screening, or longer if judged by the investigator to possibly influence the outcome of the current trial
* High daily consumption of caffeine-containing beverages (e.g. more than five cups of coffee or equivalent) with a risk of withdrawal symptoms arising during the trial that may confound the safety evaluation
* Blood donation or major blood loss (greater than equal to [≥]500 mL) within the last 8 weeks, or plasma donation with the last 4 weeks preceding the first day of IMP dosing
* Current non-smokers or light smoker with a history of long-term, heavy smoking (>10 pack-years)
* Previously dosed in this trial
* Mental incapacity or language barrier precluding adequate understanding or co-operation
* Considered by the investigator to be unsuitable to participate in the trial for any other reason

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-23 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- First Hospital Affiliated to Nanjing Medical University Jiangsu Province Hospital, Nanjing, China

REFERENCES:
- [Result] Shao F, Jiang Y, Ding S, Larsson P, Pinton P, Jonker DM. Pharmacokinetics and Safety of Follitropin Delta in Gonadotropin Down-Regulated Healthy Chinese Women. Clin Drug Investig. 2023 Jan;43(1):37-44. doi: 10.1007/s40261-022-01232-9. Epub 2022 Dec 7. PMID 36478528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at one site in China between June 2019 to December 2019.
Pre-assignment Details: A total of 133 subjects were screened, wherein, 24 subjects met the eligibility criteria and were randomized to the investigational medicinal product (IMP): 8 subjects each were exposed to Follitropin Delta (FE 999049) 12 μg, 18 μg and 24 μg, respectively. All the randomized subjects completed the trial.
Groups:
- Follitropin Delta (FE 999049) 12 μg: Participants received single subcutaneous abdominal injection of Follitropin Delta 12 μg on Day 1 of the Treatment Period.
- Follitropin Delta (FE 999049) 18 μg: Participants received single subcutaneous abdominal injection of Follitropin Delta 18 μg on Day 1 of the Treatment Period.
- Follitropin Delta (FE 999049) 24 μg: Participants received single subcutaneous abdominal injection of Follitropin Delta 24 μg on Day 1 of the Treatment Period.
Period: Overall Study
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised data from all dosed subjects. Subjects were analyzed according to the actual dose received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (6.0) | 29.5 (6.7) | 25.4 (4.6) | 27.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 24
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.2 (1.6) | 20.7 (1.9) | 22.0 (2.3) | 21.6 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve From Dosing to Infinity (AUC)
Description: Area under the concentration-time curve from dosing to infinity.
Time Frame: At -1, -0.5 and 0 hour predose, and at 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 48 hours, and 3, 4, 5, 6, 7, 8, and 9 days postdose
Population: The per-protocol (PP) analysis set comprised data from all dosed subjects except data excluded as a result of major protocol deviations. Subjects were analyzed according to the actual dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 41.3 (44.3) | 62.9 (19.7) | 83.1 (36.6)

2. Primary Outcome: Area Under the Serum Concentration-time Curve From Dosing up to Time t (AUCt)
Description: AUCt is defined as the area under the serum concentration-time curve from dosing up to time t, where t is the last time point at which the concentration is above the lower limit of quantification.
Time Frame: as for outcome 1
Population: The PP analysis set comprised data from all dosed subjects except data excluded as a result of major protocol deviations. Subjects were analyzed according to the actual dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 36.4 (38.0) | 56.6 (18.7) | 74.6 (35.9)

3. Primary Outcome: Maximum Serum Concentration Observed (Cmax)
Description: Maximum concentration observed in serum.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 0.388 (26.5) | 0.677 (29.1) | 0.825 (34.6)

4. Primary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Time of maximum observed concentration in serum.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
hour | 24.0 [16.0 to 36.0] | 24.0 [16.0 to 48.0] | 24.0 [24.0 to 28.0]

5. Primary Outcome: Apparent Total Systemic Clearance (CL/F)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 7 | 8 | 8
Liter/hour | 0.301 (46.6) | 0.286 (19.7) | 0.289 (36.6)

6. Primary Outcome: Apparent Volume of Distribution Associated With the Terminal Phase (VZ/F)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 7 | 8 | 8
Liter | 25.5 (19.5) | 20.8 (43.5) | 25.4 (31.5)

7. Primary Outcome: Terminal Elimination Half-life (t½)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 7 | 8 | 8
hour | 58.6 (47.5) | 50.5 (43.5) | 60.9 (13.6)

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Changes in Electrocardiogram (ECG)
Description: Number of participants with clinically significant abnormal changes in ECG are presented.
Time Frame: At screening, on Day -1, at 12, 24, 48 hours postdose, and at the follow-up visit (Day 11)
Population: The safety analysis set comprised data from all dosed subjects and was used for safety analysis. The safety analysis set was identical to the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 1

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Changes in Vital Signs
Description: Number of participants with clinically significant abnormal changes in vital signs (systemic blood pressures, heart rate and body temperature) are presented.
Time Frame: At screening, on Day -1, at 12, 24, 48 hours postdose, and at the follow-up visit (Day 11)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings in Laboratory Parameters
Description: Number of participants with clinically significant abnormal findings in laboratory parameters (clinical chemistry, haematology, urinalysis) are presented.
Time Frame: At screening, on Day -1 and Day 3, and at the follow-up visit (Day 11)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Clinical Chemistry | 2 | 1 | 1
  Haematology | 0 | 1 | 0
  Urinalysis | 0 | 1 | 0

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Type of AEs
Description: An AE is any untoward medical occurrence in a participant participating in a clinical trial. Number of participants with any AE (serious or non-serious) and type of AEs ( mild, moderate, severe) are presented.
Time Frame: From signed informed consent until the end-of-trial visit (Day 28)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Adverse events (AEs) | 5 | 4 | 3
  Serious AEs | 0 | 0 | 0
  Mild AEs | 5 | 3 | 3
  Moderate AEs | 0 | 1 | 0
  Severe AEs | 0 | 0 | 0

12. Secondary Outcome: Frequency of Injection Site Reactions
Description: The injection site reactions (redness, pain, itching, swelling, and bruising) will be assessed by the investigator after injection, 30 minutes, and 24 hours after administration of the IMP. Each injection site reaction will be assessed as none, mild, moderate, or severe.
Time Frame: Immediately, 30 minutes, and 24 hours after administration
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Treatment-induced Anti-follicle-stimulating Hormone (Anti-FSH) Antibodies
Time Frame: On Day 1 predose, Day 7, and Day 28
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signed informed consent until the end-of-trial visit (Day 28)
Description: A treatment-emergent AE was any AE occurring after administration of IMP and within the time of residual drug effect, or a pre-treatment AE or pre-existing medical condition that worsened in intensity after start of IMP and within the time of residual drug effect. Only treatment-emergent AEs are presented.
Arm/Group | Follitropin Delta (FE 999049) 12 μg | Follitropin Delta (FE 999049) 18 μg | Follitropin Delta (FE 999049) 24 μg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 4/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Follitropin Delta (FE 999049) 12 μg (N=8) | Follitropin Delta (FE 999049) 18 μg (N=8) | Follitropin Delta (FE 999049) 24 μg (N=8)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Smear cervix abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT04150861/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT04150861/SAP_001.pdf